CLINICAL TRIAL: NCT02840110
Title: Long-Term Follow-Up Study of Subjects Treated With an Autologous T Cell Product Expressing an Antibody-Coupled T-Cell Receptor (ACTR)
Brief Title: Long-Term Follow-Up Study of Subjects Treated With ACTR T Cell Product
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: UT-201502
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: B Cell Lymphomas; Multiple Myeloma; Solid Tumor; HER-2 Protein Overexpression
MeSH Terms: conditions — Lymphoma, B-Cell; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for replication competent retrovirus (RCR) testing
  Remaining biological samples from other protocol procedures (e.g., blood for presence of ACTR+ T cells) may also be stored, at the discretion of the sponsor, for potential future biomarker analyses of T cells, DNA, RNA, and other cells or molecules to study immunology or gene therapy.
  Optional blood, bone marrow, and tissue samples also may be collected in the event of a subject's death if an autopsy is performed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-ACTR: Subjects who have previously been treated with an ACTR T cell product
  Interventions: Other: ACTR T Cell Product

INTERVENTIONS:
Other: ACTR T Cell Product

SUMMARY:
Subjects treated with an ACTR product may participate in this long-term follow-up study after the completion of the final scheduled visit in the parent clinical study or other investigational setting, such as compassionate use, named patient Investigational New Drug application, expanded access program, or equivalent setting. No investigational product or treatment will be administered in this study. These subjects will be followed for safety monitoring on a schedule of decreasing frequency through 15 years post-ACTR treatment, in accordance with US FDA Regulatory guidance pertaining to long-term safety follow-up for study subjects receiving recombinant DNA-containing investigational products.

ELIGIBILITY:
Inclusion Criteria

* Willing to provide informed consent for participation in the study
* Received at least 1 dose of an ACTR T cell product in an investigational or other treatment setting, such as compassionate use, named patient IND, expanded access program, or equivalent settings
* Has completed study assessments and follow-up visits in the prior study or other investigational setting to the extent willing and able to do so
* Able to comply with study requirements

Exclusion Criteria

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects with disease progression after being treated with at least one dose of an ACTR T cell product in the parent study or other investigational setting
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Long-term safety of ACTR T cell product as assessed by overall survival | Total of 15 years after first receiving an ACTR T cell product
Long-term safety of ACTR T cell product as assessed by serious adverse events related to ACTR T cell product | Total of 15 years after first receiving an ACTR T cell product
Long-term safety of ACTR T cell product as assessed by Grade 3 or 4 adverse events related to ACTR T cell product | Total of 15 years after first receiving an ACTR T cell product
Long-term safety of ACTR T cell product as assessed by adverse events of special interest, regardless of grade or relatedness to the ACTR T cell product | Total of 15 years after first receiving an ACTR T cell product
ACTR T cell persistence in subjects previously treated with an ACTR T cell product | Total of 15 years after first receiving an ACTR T cell product

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sachs, MD, Study Director — Cogent Biosciences, Inc.
Locations (16):
- United States (16):
  - Banner MD Anderson, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Loyola University, Maywood, Illinois
  - Indiana Bone and Marrow Transplantation, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Baylor University Medical Center, Charles Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No